CLINICAL TRIAL: NCT01422681
Title: Extracorporeal Carbon Dioxide Removal in Patients With Severe COPD Exacerbation Failing Noninvasive Ventilation
Brief Title: Extracorporeal CO2 Removal in COPD Exacerbation
Acronym: DECOPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Marco Ranieri, MD Professor, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DECOPD1
Record Dates: First submitted 2011-08-05; First posted 2011-08-24 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: COPD Exacerbation
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DECOPD (Experimental): patients with severe COPD exacerbation on NIV treated with the minimally invasive extracorporeal carbon dioxide removal device (Decap Smart)
  Interventions: Device: minimally invasive extracorporeal carbon dioxide removal

INTERVENTIONS:
Device: minimally invasive extracorporeal carbon dioxide removal — The application of the extracorporeal carbon dioxide removal will be initiated by using a modified continuous veno-venous hemofiltration system equipped with a membrane lung with a total membrane surface of 1,35 m2 (Decap® Smart).
  Femoral vein is accessed via a double lumen catheter (14 F) inserted with the Seldinger technique and connected with the extracorporeal circuit. Blood flow is driven through the circuit by a roller nonocclusive low-flow pump (0- 450 ml/min) through a membrane lung (Euroset) that is connected to a fresh gas flow source delivering 100% oxygen at a constant rate of 8 l/min. Exiting the membrane lung, blood is driven to a hemofilter (Medica D250). The resulting plasmatic water is recirculated through the membrane lung by a peristaltic pump (0-155 ml/min).

SUMMARY:
The minimally invasive extracorporeal carbon dioxide removal may decrease the respiratory load during chronic obstructive pulmonary disease (COPD) exacerbation, reducing the need to advance the respiratory care toward invasive mechanical ventilation in patients refractory to non-invasive ventilatory support (NIV), or decreasing the need of ventilatory support in patients already invasively ventilated, thereby accelerating the weaning process.

The investigators intend to perform a multi-center experimental non randomized single arm prospective study to investigate the efficacy of the Decap Smart in reducing the intubation rate or the duration of invasive mechanical ventilation in patients with COPD treated either with NIV or invasive mechanical ventilation (IMV) for severe respiratory failure and hypercapnia. The results of the study will be compared to the data available in the literature.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* severe acute respiratory failure
* after at least two hours of continuous application of non-invasive ventilatory support (NIV):
* arterial pH ≤7.30 with an arterial pressure of CO2 (PaCO2) >20% of the baseline value and one of the following:
* respiratory rate ≥30 breaths/min;
* use of accessory muscles or paradoxical abdominal movements

Exclusion Criteria:

* failure to obtain consent
* hemodynamic instability (MAP < 60 mmHg) despite infusion of vasoactive drugs
* contraindications to the administration of i.v. heparin (heparin induced thrombocytopenia, hemorrhage, etc.)
* body weight >120 kg
* contraindication to continuation of active treatment (DNR)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
number of patients treated with the Decap Smart failing NIV and therefore needing endotracheal intubation | 1 month

SECONDARY OUTCOMES:
Adverse events | 1 month
Hospital length of stay | 18 months
ICU length of stay | 18 months
Hospital mortality | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: V. Marco Ranieri, MD, Study Director — University of Turin, Italy
Locations (1):
- University of Turin, Department of Anesthesia and Intensive Care Medicine, Turin, Italy, Italy

REFERENCES:
- [Derived] Del Sorbo L, Pisani L, Filippini C, Fanelli V, Fasano L, Terragni P, Dell'Amore A, Urbino R, Mascia L, Evangelista A, Antro C, D'Amato R, Sucre MJ, Simonetti U, Persico P, Nava S, Ranieri VM. Extracorporeal Co2 removal in hypercapnic patients at risk of noninvasive ventilation failure: a matched cohort study with historical control. Crit Care Med. 2015 Jan;43(1):120-7. doi: 10.1097/CCM.0000000000000607. PMID 25230375